CLINICAL TRIAL: NCT03021083
Title: Evaluating the Feasibility of Using Transdermal Patient-controlled Fentanyl After Spinal Fusions
Brief Title: IONSYS Feasibility Study
Acronym: IONSYS Pilot
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Contract not reached with sponsor
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-803
Record Dates: First submitted 2016-12-16; First posted 2017-01-13 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Spinal Injury
Keywords: Lumbar multi-level fusions; Patient Controlled Analgesia; Fentanyl; Opioid Analgesia
MeSH Terms: conditions — Spinal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- IONSYS Administration (Experimental): Patients who have elective multi-level spinal fusions under general anesthesia (who do not receive methadone) will be enrolled. In addition, all patients will receive Pepcid 20 mg, dexamethasone 10 mg, and ondansetron 4 mg.
  When patients will arrive in the post anesthesia care unit (PACU), pain will initially be controlled with IV hydromorphone to achieve an NRS score of 3 or less. Once transferred to the step down unit (SDU), the IONSYS patch will be applied. IONSYS should be utilized when they have pain, but rescue analgesia will be available. If severe pain continues, the chronic pain service will be consulted, to potentially change the medications.
  Patients will be assessed for pain at rest and with PT in the AM and PM of POD 1 and POD 2. The IONSYS system will be discontinued after 48 hours, and a total dose of fentanyl received per 24 hours will be recorded. PT milestones for discharge will be assessed on the afternoon of POD 1 and POD 2.
  Interventions: Device: IONSYS Patch

INTERVENTIONS:
Device: IONSYS Patch — Patient controlled transdermal fentanyl patch, IONSYS, applied to patient in place of a PCA.
  Other Names: Patient Controlled Transdermal Fentanyl Patch

SUMMARY:
The treatment of postoperative pain continues to be a challenge after posterior spinal fusions. There is considerable evidence demonstrating that a multi-modality approach including patient controlled analgesia (PCA) with opioids for postoperative pain management compared to conventional opioid analgesia provides a greater analgesic effect even when the amount of opioids consumed is similar between both groups. However, the PCA modality is often discontinued prior to all the patients' pain needs being met. The IONSYS system uses the concept of PCA-delivered narcotics and may be used for postoperative pain management.

DETAILED DESCRIPTION:
Following posterior spinal fusions, many patients are treated with analgesics or other modalities for prolonged periods before choosing the surgical alternative. In addition, the narcotic-based anesthetic required for the procedure may induce postoperative hyperalgesia (1). Inadequate treatment of this pain can result in prolonged hospitalization, cardiopulmonary complications, and poor surgical outcome (2).

Pain during the immediate postoperative period is usually managed with IV narcotic PCA and then transitioned to a combination of long-acting and short-acting oral analgesics. Because of the requirement for continuous carrier fluid infusion, cumbersome pump technology restricting mobility and supervision by a dedicated pain team to control programming of the pump, the PCA modality is often discontinued prior to all the patients' pain needs being met.

The investigators' most recent study evaluated the addition of pregabalin to the pain regimen after spinal fusions. The study found that after the removal of the PCA modality, these patients had considerable pain during physical therapy (PT), and their pain was not improved with the addition of pregabalin.

The IONSYS system might alleviate some of the problems encountered with conventional PCA systems (3,4). The system is an iontophoretic transdermal (needleless) system preprogrammed to deliver upon activation 40 mcg fentanyl over a 10-minute period, with up to 6 doses per hour. The system performs for 24 hours. The drug is embedded in a matrix gel and is only delivered when a current is propagated between the two poles of the system. Other than the usual narcotic side effects, the only specific side effect is a local dermatological reaction to the patch (5% had a rash, which cleared after removal). The system was designed with fentanyl, since hydromorphone cannot be incorporated in this type of matrix. Unlike hydromorphone, fentanyl is quick acting and doesn't hang around. The in-house chronic pain service currently puts many of their patients on IV fentanyl, because of the belief that it works when they have pain but is quickly metabolized.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-70 years old undergoing elective multi-level lumbar-sacral posterior spinal fusions

Exclusion Criteria:

* Chronic pain patients taking more than 20-mg equivalents of oxycodone daily
* Allergy to either hydromorphone or fentanyl
* Other chronic orthopedic pain complaints, which will confound the results of the study
* Issues with cognitive ability

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of IONSYS system | Day 2 following surgery for each patient
  1. Nursing assessment regarding the ease of setup and initiation of the IONSYS system (With regard to setup and initiation of the IONSYS, on a scale of 0-10, where 0=worst and 10=best, how would the nurse rate the system?). This will be given to the nurse who sets up the device on DOS, and nurse who sets up the device on POD 1, and the day nurse on POD 2. An average score of 7 will be considered feasible.
NRS Pain Scores | Day 1 following surgery for each patient
  1. NRS pain (0-10 scale) on first day after surgery (POD 1) during the afternoon session of PT. In a previous study on similar patients with IV PCA, we recorded mean pain scores of 4.6 during PT. Adequate pain control is delineated as NRS ≤ 3

SECONDARY OUTCOMES:
Day of eligibility for discharge, | Up to 1 week after surgery
  1. Day of eligibility for discharge, as assessed by a physical therapist's observation of a patient's ability to walk at least 20 feet and climb 4 stairs. Will be delineated as either AM or PM on a day following surgery, since PT is conducted twice daily.
A Oswestry Back Pain Disability Index questionnaire | 6 weeks after surgery at the Post-Op Office Visit
  An Oswestry Back Pain Disability Index questionnaire will be conducted at the first postoperative office visit to assess whether improved pain control in the hospital had an effect on the post-discharge recovery of the patient.
Level of Sedation | POD1
  Level of sedation, as assessed by PT starting on POD1 at the initiation of PT using the University of Michigan sedation scale: (1) awake and alert; (2) minimally sedated; (3) moderately sedated; (4) deeply sedated; (5) unarousable
Presence of Nausea of Vomiting | POD1 and POD2 after surgery
  Assess whether the patient has post-operative nausea and vomiting (PONV)
Satisfaction Survey | Up to 1 week
  A satisfaction survey will be conducted prior to discharge from the hospital. It will include the following questions: (1) Was the patient's pain adequately treated? (Y/N); (2) What was the patient's worst pain level after surgery? (0-10 scale); (3) Was the IONSYS device explained? (Y/N); (4) Did the patient have side effects to the IONSYS? (Y/N); (5) Was the patient able to perform PT? (Y/N); (6) Overall satisfaction with IONSYS device (0-10 scale; 0=not satisfied; 10=most satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Urban, M.D., Principal Investigator — Hospital for Special Surgery, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. PMID 24829420
- [Background] White PF. The changing role of non-opioid analgesic techniques in the management of postoperative pain. Anesth Analg. 2005 Nov;101(5 Suppl):S5-S22. doi: 10.1213/01.ANE.0000177099.28914.A7. PMID 16334489
- [Background] Scott LJ. Fentanyl Iontophoretic Transdermal System: A Review in Acute Postoperative Pain. Clin Drug Investig. 2016 Apr;36(4):321-30. doi: 10.1007/s40261-016-0387-x. PMID 26968174
- [Background] Mayes S, Ferrone M. Fentanyl HCl patient-controlled iontophoretic transdermal system for the management of acute postoperative pain. Ann Pharmacother. 2006 Dec;40(12):2178-86. doi: 10.1345/aph.1H135. PMID 17164395